CLINICAL TRIAL: NCT02774317
Title: A Pilot Study to Compare the Use of Fresh Frozen Plasma With 24-Hour Plasma in Babies Up to Age Six Months
Brief Title: Pilot Study to Compare Fresh Frozen Plasma With 24-Hour Plasma in Babies Up to Age Six Months
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The clinical team couldn't recruit patients who met the criteria for enrollment
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB15-0795
Record Dates: First submitted 2015-12-01; First posted 2016-05-17 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Blood Coagulation Disorders
MeSH Terms: conditions — Blood Coagulation Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FFP (Active Comparator): Patients receive FFP as clinically indicated (INR 1.5 or more)
  Interventions: Biological: Plasma
- FP24 (Experimental): Patients receive FP24 as clinically indicated (INR 1.5 or more)
  Interventions: Biological: Plasma

INTERVENTIONS:
Biological: Plasma — FFP (plasma frozen within 8 hrs of collection) or FP24 (plasma frozen within 24 hrs of collection)

SUMMARY:
With the advent of measures to try to decrease the incidence of transfusion-related acute lung injury (TRALI), the Blood Bank industry is attempting to avoid collection of plasma from female donors who have been pregnant in order to reduce the transfusion of plasma that may contain HLA antibodies. This has led to a decrease in the number of donors available for the production of fresh frozen plasma (FFP). Per Blood Bank regulatory standards in the United States, FFP must be frozen within 8 hours of collection. Plasma that is frozen within 24 hours of collection is called FP24, and it is produced when whole blood cannot be processed within the 8-hour time period for the generation of FFP. Studies of coagulation factors in FFP and FP24 have shown that coagulation factor activities are adequate to maintain hemostasis in both products. Many hospitals are using FFP and FP24 interchangeably in adults, and occasional hospitals are using these products interchangeably in neonates. However, studies concerning the use of FP24 in neonates have not been performed.

The investigators propose a single center prospective pilot study comparing the clinical efficacy of FFP vs. FP24 in 50 nonsurgical neonates and babies up to age 6 months requiring plasma for an International Normalization Ratio (INR) of 1.5 or more.

This protocol describes a pilot study to compare the use of FFP with FP24 in nonsurgical neonates. Use of plasma in these cases is mostly for patients with perinatal hypoxia or necrotizing enterocolitis and an INR of 1.5 or more. Transfusion of plasma (10 to 15 ml/kg) is performed for these patients approximately every 8, 12, or 24 hours, as deemed indicated by the patient's clinicians, and monitored with prothrombin time (PT), partial thromboplastin time (PTT), and INR.

DETAILED DESCRIPTION:
Half the patients will be randomized by the Blood Bank to receive FFP, the other half FP24. All patients will be monitored in the usual way, with careful clinical observation and with PT/PTT/INR, to be drawn once in 12 or 24 hours based on clinical necessity. If a patient needs additional transfusions, the same type of product will be administered for each episode.

ELIGIBILITY:
Inclusion Criteria:

* Nonsurgical neonates and babies up to age 6 months with INR 1.5 or more who are deemed clinically to need plasma infusion.

Exclusion Criteria:

* Patients who are being prepared for surgery, or during or after surgery.
* Patients with congenital anomalies, chromosomal anomalies, or heart defects.
* Patients whose parents refuse to consent.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-10 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Number of neonates with corrected International Normalization Ratio (INR)upon transfusion with plasma frozen within 24 hours of collection (FP24) | 24 hrs
  The investigators will compare fresh frozen plasma (FFP) with FP24 in correcting INR in 50 nonsurgical neonates

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No